CLINICAL TRIAL: NCT03646357
Title: BEtablocker Treatment After Acute Myocardial Infarction in Patients Without Reduced Left Ventricular Systolic Function (BETAMI)
Brief Title: BEtablocker Treatment After Acute Myocardial Infarction in Patients Without Reduced Left Ventricular Systolic Function
Acronym: BETAMI
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Vestre Viken Hospital Trust (Other); The Hospital of Vestfold (Other); University of Oslo (Other); Helse Stavanger HF (Other Government); Haukeland University Hospital (Other); St. Olavs Hospital (Other); University Hospital of North Norway (Other); Sorlandet Hospital HF (Other Government); Norwegian University of Science and Technology (Other); Sykehuset Innlandet HF (Other); Nordlandssykehuset HF (Other); Lovisenberg Diakonale Hospital (Other); Diakonhjemmet Hospital (Other); Ostfold Hospital Trust (Other)
Responsible Party: Principal Investigator, Dan Atar, Professor of Cardiology, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-000590-75
Record Dates: First submitted 2018-05-14; First posted 2018-08-24 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Acute Myocardial Infarction; Non-ST Elevation Myocardial Infarction; ST Elevation Myocardial Infarction
Keywords: Infarction; Myocardial Infarction; ST Elevation Myocardial Infarction; Non-ST Elevated Myocardial Infarction; Ischemia; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Metoprolol; Bisoprolol; Betablocker; Anti-Arrhythmia Agents; Physiological Effects of Drugs; Beta-blocker; Beta blocker
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction; Infarction; Myocardial Infarction; Ischemia; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: PROBE - prospective, randomized, open blinded end-point
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Betablocker (Active Comparator): Patients receiving a betablocker. Any other treatment or management is to be given as per usual care.
  Interventions: Drug: Betablocker
- Non-Betablocker (Experimental): No betablocker is given to this arm. Any other treatment or management is to be given as per usual care.
  Interventions: Other: Non-betablocker

INTERVENTIONS:
Other: Non-betablocker — No betablocker will be administered. Patients randomized to no beta-blockade will be discouraged to use beta-blockade as long as there is no other indication than strictly secondary prevention after myocardial infarction. Any other treatment or management is to be given as per usual care.
  Arms: Non-Betablocker
Drug: Betablocker — A betablocker will be administered. To reflect contemporary management, for which this study is designed to test, there will not be a defined minimum dosage. The type and dose of BB will be left at the discretion of the PI. Generic drug and accepted dosages will be:
  * Metoprolol succinate up to a total dose of 200mg daily
  * Bisoprolol up to a total dose of 10mg daily
  * Carvedilol up to a total dose of 50mg daily
  The treating physician will be encouraged to aim for an equipotent dose of 100 mg metoprolol succinate or higher. Any other treatment or management is to be given as per usual care.
  Arms: Betablocker

SUMMARY:
The study aims to investigate whether oral betablocker (BB) therapy is superior to no such treatment following an acute myocardial infarction (AMI).

DETAILED DESCRIPTION:
This is a prospective, randomized, open blinded end-point (PROBE) study. Patients with AMI will be randomized 1-8 days following PCI or thrombolysis, and allocated to either prescription of a BB or to no such prescription. Subjects will be followed up for at least 6 months (median 3 years) with respect to the primary and secondary endpoints. The primary end point, the key secondary end points, and most other secondary end points will be analysed and published jointly with data from the 'Danish Trial of Beta-blocker therapy after myocardial infarction without heart failure' (DANBLOCK) (NCT 03778554) (please see below).

The primary objective is to test whether oral BB therapy reduces the risk of all-cause death, recurrent MI, incident heart failure, unplanned coronary revascularization, ischemic stroke, or malignant ventricular arrhythmia including resuscitated cardiac arrest of cardiac origin compared to no such therapy, in patients with AMI treated with PCI or thrombolysis without reduced LVEF.

The key secondary objectives (planned for the main study) are:

* To study whether oral BB therapy reduces the risk of each of the components of the primary end-point separately, compared to no such therapy
* To assess clinical outcomes linked BB therapy in the following subgroups: age (tertiles< 70 years vs. ≥70 years), gender sex (men vs. women), country (Denmark vs Norway), BB dosage tertiles (dosage at randomization (<50 mg vs. ≥50 mg), hypertension (yes vs. no), diabetes (yes vs. no), diabetes (yes vs no), type of MI (STEMI vs. NSTEMI), and LVEF subgroups (preserved LVEF: ≥50% vs. mid-range LVEF: 40-49%).
* To study whether oral BB therapy increases the risk of hospitalization for second or third-degree atrioventricular block or implantation of pacemaker.
* To describe BB dosage and adherence at six months following randomization obtained from the national prescription registries
* To assess study safety

Other secondary objectives (for joint BETAMI-DANBLOCK sub-studies) are:

* To study whether oral BB therapy reduces the risk of cardiovascular death compared to no such therapy
* To study whether oral BB therapy reduces the risk of stable and unstable angina compared to no such therapy
* To study whether oral BB therapy reduces the risk of atrial fibrillation, atrial flutter or other atrial tachyarrhythmias compared to no such therapy
* To study whether oral BB therapy increases the risk of hospitalization for bradycardia or syncope.
* To study whether oral BB therapy increases the risk of hospitalization for chronic obstructive pulmonary disease, asthma or peripheral artery disease.
* To study whether oral BB therapy affects the following patient related outcomes:

quality of life, angina, dyspnoea, anxiety, depression, sexual dysfunction or sleep disorders

* To describe long term BB adherence obtained from the national prescription registries
* To study sociodemographic, clinical, and psychosocial characteristics (PROMS and clinical data) between the two study arms and in the total sample
* To conduct cost-utility analysis in relation to quality of life and a health economic evaluation including drug use, health care utilization, employment, income, and benefit take-up

Exploratory objectives (based on BETAMI data, only):

* To study the proportion and predictors of non-adherence with BB, statins and other cardiovascular drugs assessed by direct methods quantifying drug concentrations in blood
* Identify pharmacokinetic, pharmacogenetic and pharmacodynamic markers associated with side-effects and suboptimal response to treatment with cardiovascular drugs

The primary study end-points will be obtained through linkage to the Norwegian Cardiovascular Disease Registry and The Norwegian Population Registry (Folkeregisteret)

Secondary endpoints will be obtained by linkage to the following national registries: The Norwegian Population Registry (Folkeregisteret), the Cause of Death Registry, the Norwegian Patient Registry, the Norwegian Cardiovascular Disease Registry, the Norwegian Prescription Database, the Norwegian registry for income, the FD-Trygd database (social security micro data for research) and the Control and payment of reimbursements to health service providers (KUHR) database. Further by collecting self-reported questionnaires and a clinical examination with blood sample collection.

Primary safety endpoints:

• To describe the composite endpoint of malignant ventricular arrhythmias including resuscitated cardiac arrest of cardiac origin, incident heart failure, new MI or all-cause death at 30 days after randomization collected from i. direct telephone contact with the patient and from hospital medical records, ii. linkage to the Norwegian Cardiovascular Disease Registry and The Norwegian Population Registry at study end.

Other safety endpoints:

* To describe all-cause death at study end
* To describe Suspected Unexpected Serious Adverse Reaction (SUSARs) during the follow-up period from the study database (continously reported by local investigators).

Rationale for combining data from the BETAMI study with the DANBLOCK (NCT03778554) study from Denmark: The trials have similar designs, only minor differences in study entry criteria, and were, from the very beginning, coordinated with the aim of conducting sub-studies on pooled data. However, the inclusion- and event rates have been lower than expected in both studies. To enhance feasibility, the final decision was made from both Steering Committees in May 2021 to combine the trials and publish initial results jointly. BETAMI and DANBLOCK will remain separate trials until the end of follow-up, where data from the trials will be combined and main results published together.

Sample size: A total of approximately 2900 patients from BETAMI will be recruited and randomized 1:1 to BB treatment (type and dosage according to treating physician) or no BB treatment within 8 days of MI. The study is event driven and a power calculation for the combined DANBLOCK-BETAMI trial has been performed in which 950 events will provide a power of 80% to detect a true treatment effect equal to a hazard ratio of 1.2 for no beta-blocker therapy. Follow-up: Patients will be followed from the randomization date until end of follow-up. The last patient included will be followed for a minimum of 6 months. Estimated mean (non) treatment duration is 3 (0.5-6) years.

Post-trial objective:

• To perform a joint analysis of the data from BETAMI-DANBLOCK with the REDUCE (NCT03278509), CAPITAL-RCT (NCT01155635) and REBOOT (NCT03596385) trials. This analysis will comprise approximately 19000 patients, giving increased power and precision for clinical decisions on both primary and secondary endpoints.

ELIGIBILITY:
Inclusion Criteria

To be eligible for inclusion in the study, subjects must fulfill the following criteria at inclusion:

* 18 years or older
* Diagnosed with an acute MI type I according to the "Universal Definition of MI" (Defined as a detection of a rise and/or fall of cardiac biomarker value, preferably troponin, with at least one value above the 99th percentile upper reference limit and with at least one of the following; a) symptoms of ischemia, b) new or presumed new significant ST-segment-T wave changes or new left bundle branch block, c) development of pathological Q waves, d) imaging evidence of new loss of viable myocardium or e) identification of an intracoronary thrombus by coronary angiogram)
* Must have been treated with PCI or thrombolysis during current hospitalization
* Signed informed consent and expected cooperation of the patient according to ICH/GCP and national/local regulations
* Have a national personal identification number and not be expected to emigrate during study

Exclusion Criteria

Study subjects must not meet any of the following criteria:

* Having a condition where betablocker-therapy is required, including but not limited to:

  * Arrhythmias
  * Hypertension
  * Cardiomyopathies
  * Clinical diagnosis of heart failure
  * LVEF < 40% by echocardiography (by measurement and not only visual assessment for STEMI patients)
  * Left ventricular akinesia in ≥ 3 segments regardless of the LVEF
* Contraindications to betablocker-therapy, including but not limited to:

  * Bradyarrhythmias
  * Hypotension
  * Severe peripheral artery disease
  * Previously known side-effects causing withdrawal
  * Severe chronic obstructive pulmonary disease
  * • Women of childbearing potential (a woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile)
* Known hypersensitivity to any ingredient of the IMP
* Other, according to the responsible investigator
* End-stage somatic disease with short life expectancy, dementia, psychosis and other conditions could put the subject at significant risk, confound the study results, interfere significantly with the subject participation in the study, or rendering informed consent unfeasible

Previous treatment with a betablocker is not an exclusion criterion for enrollment into the BETAMI study. Enrolled patients can participate in any other study that does not directly alter the effect betablocker treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2895 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2035-12-10 (Estimated)

PRIMARY OUTCOMES:
A composite of death of any cause, recurrent myocardial infarction, incident heart failure, coronary revascularization, ischemic stroke, malignant ventricular arrhythmia including resuscitated cardiac arrest of cardiac origin | 6 months (minimum) to 6 years (maximum)
  Incidence of combined endpoint from randomization. Estimated maximal follow-up for each patient for this outcome is 6 months to 6 years

SECONDARY OUTCOMES:
Recurrent MI | 6 months (minimum) to 6 years (maximum)
  Time to recurrent MI from randomization. Estimated maximal follow-up for each patient for this outcome is 6 months to 6 years
All-cause death | 6 months (minimum) to 6 years (maximum)
  Time to a-cause Death from randomization. Estimated maximal follow-up for each patient for this outcome is 6 months to 6 years
Malignant ventricular arrhythmias including resuscitated cardiac arrest of cardiac origin | 6 months (minimum) to 6 years (maximum)
  Time to malignant ventricular arrhythmia including resuscitated cardiac arrest of cardiac origin from randomization. Estimated maximal follow-up for each patient for this outcome is 6 months to 6 years
Hospitalization or outpatient consultation for incident heart failure | 6 months (minimum) to 6 years (maximum)
  Time to hospitalization or outpatient consultation for heart failure from randomization. Estimated maximal follow-up for each patient for this outcome is 6 months to 6 years
Unplanned coronary revascularization | 6 months (minimum) to 6 years (maximum)
  Time to unplanned coronary revascularization from randomization. Estimated maximal follow-up for each patient for this outcome is 6 months to 6 years
Ischemic stroke | 6 months (minimum) to 6 years (maximum)
  Time to ischemic stroke from randomization. Estimated maximal follow-up for each patient for this outcome is 6 months to 6 years
Cardiovascular death | 6 months (minimum) to 6 years (maximum)
  Time to cardiovascular death from randomization. Estimated maximal follow-up for each patient for this outcome is 6 months to 6 years
Hospitalization for stable and unstable angina | 6 months (minimum) to 6 years (maximum)
  Time to hospitalization for stable and unstable angina from randomization. Estimated maximal follow-up for each patient for this outcome is 6 months to 6 years
Hospitalization for atrial fibrillation, atrial flutter or other atrial tachyarrhythmias | 6 months (minimum) to 6 years (maximum)
  Time to hospitalization for atrial fibrillation, atrial flutter or other atrial tachyarrhythmias from randomization. Estimated maximal follow-up for each patient for this outcome is 6 months to 6 years
Hospitalization for bradycardia, syncope or implantation of pacemaker | 6 months (minimum) to 6 years (maximum)
  Time to hospitalization for bradycardia, syncope or implantation of pacemaker from randomization. Estimated maximal follow-up for each patient for this outcome I 6 months to 6 years
Hospitalization for chronic obstructive pulmonary disease, asthma or peripheral artery disease | 6 months (minimum) to 6 years (maximum)
  Time to hospitalization for chronic obstructive pulmonary disease, asthma or peripheral artery disease from randomization. Estimated maximal follow-up for each patient for this outcome is 6 months to 6 years
Angina symptoms | Through self-report questionnaires administered at inclusion, 30 days, 3,6 and 18 months
  Canadian Cardiovascular Society (CCS) grading of angina pectoris.
Health-related quality of life | Through self-report questionnaires administered at inclusion, 30 days, 3,6 and 18 months
  Health-related quality of life measured by the Short Form (SF) 12
Measures of depression and anxiety | Through self-report questionnaires administered at inclusion, 30 days, 3,6 and 18 months
  HADS (Hospital Anxiety and Depression Scale)
Measures of sexual dysfunction | Through self-report questionnaires administered at inclusion, 30 days, 3,6 and 18 months
  The International Index of Erectile Function (IIEF) and Female Sexual Function Index (FSFI)
Measures of sleep disorders | Through self-report questionnaires administered at inclusion, 30 days, 3,6 and 18 months
  Bergen insomnia Scale
Measures of sleep disorders | Through self-report questionnaires administered at inclusion, 30 days, 3,6 and 18 months
  Bergen insomnia Scale and sleep duration
Measures of Nightmare Frequency | Through self-report questionnaires administered at inclusion, 30 days, 3,6 and 18 months
  Nightmare Frequency Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dan Atar, MD Prof, Study Chair — Oslo University Hospital
Locations (20):
- Norway (20):
  - Sørlandet Sykehus, Arendal
  - Haukeland Universitetssykehus, Bergen
  - Nordlandssykehuset HF Bodø, Bodø
  - Drammen Hospital, Drammen
  - Sykehuset Østfold Kalnes, Fredrikstad
  - Sykehuset Innlandet HF, Gjøvik Sykehus, Gjøvik
  - Sykehuset Innlandet Hamar, Hamar
  - Vestre Viken HF, Ringerike Sykehus, Hønefoss
  - Sykehuset Innlandet Lillehammer, Lillehammer
  - AHUS, Lørenskog
  - LHL Gardermoen, Lørenskog
  - Diakonhjemmet Sykehus, Oslo
  - Lovisenberg Diakonale Sykehus, Oslo
  - Oslo University Hospital Rikshospitalet, Dept.of Cardiology, Oslo
  - Oslo University Hospital Ullevaal, Dept. of Cardiology, Oslo
  - Vestre Viken HF, Bærum Sykehus, Sandvika
  - Stavanger Universitetssjukehus, Stavanger
  - Universitetssykehuset Nord-Norge, UNN, Tromsø
  - St. Olavs University Hospital, Trondheim
  - Vestfold hospital, Tønsberg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Munkhaugen J, Kristensen AMD, Halvorsen S, Holmager T, Olsen MH, Bakken A, Sehested TSG, Ruddox V, Maeng M, Vikenes K, Jensen SE, Steigen T, Lambrechtsen J, Jortveit J, Bovin A, Schirmer H, Christiansen MK, Wiseth R, Mikkelsen D, Larsen AI, Lyngby Kjaergaard C, Andresen K, Gustafsson I, Tuseth V, Larsen ML, Deeg PS, Veien K, Bohmer E, Botker HE, Brattrud AO, Bronnum-Schou J, Pettersen AR, Bang LE, Oie E, Engstrom T, Borg EB, Kristensen K, Nymo SH, Gislason G, Vethe NT, Abdulla JAM, Dammen T, Mouridsen MR, Bendz B, Bertelsen MLN, Hove JD, Schierbeck L, Snoer M, Davidsen C, Egholm G, Thomsen KK, Jadou G, Poenaru M, Krarup NT, Bottcher M, Staehr PB, Zwisler AD, Edvardsen T, Torp-Pedersen C, Otterstad JE, Lange T, Fagerland MW, Atar D, Prescott E; BETAMI-DANBLOCK Investigators. Beta-Blockers after Myocardial Infarction in Patients without Heart Failure. N Engl J Med. 2025 Nov 13;393(19):1901-1911. doi: 10.1056/NEJMoa2505985. Epub 2025 Aug 30. PMID 40888716
- [Derived] Granger CB, Pocock SJ, Gersh BJ. The need for new clinical trials of old cardiovascular drugs. Nat Rev Cardiol. 2023 Feb;20(2):71-72. doi: 10.1038/s41569-022-00819-1. No abstract available. PMID 36526898

DOCUMENTS (2):
  • Study Protocol (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT03646357/Prot_002.pdf
  • Statistical Analysis Plan (2025-03-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT03646357/SAP_004.pdf